CLINICAL TRIAL: NCT01187537
Title: Effects of Continuous Femoral Nerve Block Versus Single-Injection Femoral Nerve Block With Intravenous Patient Controlled Analgesia Versus Intravenous Patient Controlled Analgesia on Knee Pain and Function After Total Knee Replacement
Brief Title: Effects of Continuous Nerve Block vs Single Injection Block With PCA vs PCA on Pain and Function After Knee Replacement
Acronym: PCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Chan Ee Yuee, Dr, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIG/09052
Record Dates: First submitted 2010-08-22; First posted 2010-08-24 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2010-08

CONDITIONS: Pain
Keywords: Knee Replacement; Analgesia; Analgesics; Nerve blocks; Recovery of functions; Post operative analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuous Femoral Nerve Block (Experimental)
  Interventions: Procedure: Continuous Femoral Nerve Block
- Single-Inj Nerve Block with IV PCA (Active Comparator)
  Interventions: Procedure: Continuous Femoral Nerve Block
- IV PCA (Active Comparator)
  Interventions: Procedure: Continuous Femoral Nerve Block

INTERVENTIONS:
Procedure: Continuous Femoral Nerve Block — 20mls of 0.25% Bupivacaine with 1/400,000 adrenaline (2.5mcg/ml) If catheter localized to < 1.0mA, 0.1mS with patella twitch, start Bupivacaine 0.125% 4ml/hr. If unable to get twitch through catheter in final location or twitch at current ≥ 1.0m/A, start Bupivacaine 0.125% 6ml/hr.
  Other Names: Bupivacaine

SUMMARY:
The purpose of this study is to compare the effectiveness of three analgesia techniques on pain relief and functional recovery after knee replacement: continuous femoral nerve block vs single-injection femoral nerve block with intravenous patient controlled analgesia vs intravenous patient controlled analgesia.

DETAILED DESCRIPTION:
Primary Outcome Measures:

* Incidence of patients with significant pain on movement on day 1 post surgery
* Range of knee flexion

Secondary Outcome Measures:

* Pain intensity (rest/movement)
* Functional recovery
* Knee Injury and Osteoarthritis Score
* Side effects/ Adverse outcomes
* SF12 Quality of Life Questionnaire
* Length of stay

ELIGIBILITY:
Inclusion Criteria:

* 40 years and above
* Osteoarthritis
* Primary unilateral total knee replacement
* No other lower extremity joint disease
* ASA I-III
* Body mass index < 35
* No severe cardiac or pulmonary diseases
* No chronic narcotic therapy or illicit drug use
* Mentally competent to understand study procedures and use of pain scales
* Able to provide informed consent

Exclusion Criteria:

* Any cause for knee replacement other than osteoarthritis
* Total knee revision
* Any contraindication for femoral block
* Abnormal coagulation studies
* Thrombocytopenia less than 100,000/cc
* Known hepatic or renal insufficiency
* Neurological disease involving lower extremities
* Major surgery during the last 2 weeks pre-operatively
* History of allergy to study medications
* History of post-operative bleeding over 2000 cc/24 hours
* History of opioid or alcohol abuse
* Currently taking or has taken opioid > 30 consecutive days of daily use at a daily dose > 15mg morphine, within the past 2 weeks prior to surgery
* Previously has not responded to opioid analgesics for treatment of pain
* Pregnancy or breastfeeding

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with significant pain on movement on day 1 post surgery | Post op day 1

SECONDARY OUTCOMES:
Functional recovery | During hospitalization, week 2, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ee Yuee Chan, Principal Investigator — Tan Tock Seng Hospital; Nelson Chua, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Chan EY, Teo YH, Assam PN, Fransen M. Functional discharge readiness and mobility following total knee arthroplasty for osteoarthritis: a comparison of analgesic techniques. Arthritis Care Res (Hoboken). 2014 Nov;66(11):1688-94. doi: 10.1002/acr.22361. PMID 24782108